CLINICAL TRIAL: NCT06852469
Title: Individualized Computational Assessment of the Effects of GABA Receptor Modulation in Posttraumatic Stress Disorder
Brief Title: Computational Assessment of GABA Receptor Modulation in PTSD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: MHBP-009-24S
Record Dates: First submitted 2025-02-21; First posted 2025-02-28 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Arousal; gamma-Aminobutyric Acid; Lorazepam; Neuroimaging; Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Lorazepam; Tablets

STUDY DESIGN:
Intervention Model Description: Each included participant will be administered a dose of lorazepam 1 mg and placebo in a crossover design, with the order of lorazepam and placebo determined in double-blind, randomized fashion (using a randomly permuted block design), with a one-week washout period
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Assignment will be balanced using a randomly permuted block design. Medication will be prepared and labeled by a research pharmacist not otherwise involved in the study, and both participant and study personnel will be blinded to the study drug being administered. In case of medical emergency, unblinding can be performed. The pharmacy will blind drug and placebo through identical encapsulation. Placebo will match the study drug in mode of administration, color, size, and taste.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lorazepam 1 mg, then placebo (Experimental): Participants will first receive a single dose of lorazepam 1 mg on the first testing session. After a 1 week washout period, participants will then receive a single dose of placebo on the second testing session.
  Interventions: Drug: Lorazepam 1 mg tablet; Drug: Placebo tablet
- Placebo, then lorazepam 1 mg (Experimental): Participants will first receive a single dose of placebo on the first testing session. After a 1 week washout period, participants will then receive a single dose of lorazepam 1 mg on the second testing session.
  Interventions: Drug: Lorazepam 1 mg tablet; Drug: Placebo tablet

INTERVENTIONS:
Drug: Lorazepam 1 mg tablet — Lorazepam is an oral medication which is FDA approved to treat anxiety.
  Other Names: Ativan
Drug: Placebo tablet — Placebo will match the study drug in mode of administration, color, size, and taste.

SUMMARY:
A substantial majority of Veterans with posttraumatic stress disorder (PTSD) continue to suffer even with the best current medications. Progress in developing more effective medications is hampered by the substantial variability within Veterans with PTSD, meaning the most effective medication likely varies from individual to individual. New scientific tools to help identify distinct subgroups of Veterans with PTSD who are likely to respond to specific medications could help improve treatment in this population. Research has indicated that a specific subgroup of Veterans with PTSD with a high level of anxious arousal may benefit from medications which boost signaling of the neurotransmitter gamma-aminobutyric acid (GABA). This project aims to validate a clinical test to identify these individuals using new computational and neuroimaging methods combined with the medication lorazepam, a positive GABA modulator. The ultimate goal is to use these methods in future clinical trials of new medications to target the best treatments to individual Veterans with PTSD.

DETAILED DESCRIPTION:
Heterogeneity in Veterans with PTSD has been identified as a major obstacle in developing effective treatments for this population. Research suggests that a PTSD subgroup characterized by elevated arousal, relative to general negative affect, may benefit from novel medications that positively modulate inhibitory gamma aminobutyric acid (GABA) signaling. An objective, functional phenotypic marker for this subgroup could therefore enable targeted treatment and improve clinical outcomes. The investigators propose a computational goal-directed control paradigm as a novel clinical assessment based on the premise that a reduction in dynamic inhibition, regulated by GABA signaling, can serve as a specific, objective phenotypic target in a high arousal PTSD (HA-PTSD) subgroup. This study will leverage: 1) a single dose of a benzodiazepine as an acute GABA receptor modulator for phenotypic target validation rather than treatment purposes; 2) a novel computational control modeling strategy to precisely measure the effect of GABA receptor modulation on dynamic inhibition; 3) functional neuroimaging to assess specific neural mechanisms of GABAergic influence on dynamic inhibition.

The investigators have developed the rapid assessment of motor processing (RAMP) paradigm, a computational goal-directed control task which enables precise estimation of a dynamic inhibition parameter. Compared to other behavioral measures, dynamic inhibition exhibits excellent measurement reliability. Dynamic inhibition is negatively associated with subjective fear, and this relationship persists after controlling for general negative affect. Critically, dynamic inhibition is lower in an HA-PTSD subgroup (with high residual fear, controlling for negative affect) compared to both a low arousal PTSD (LA-PTSD) subgroup and healthy controls (HC). Dynamic inhibition is also associated with structure and function in arousal-related regions such as dorsal anterior cingulate cortex (dACC) and insula.

Benzodiazepines are robust positive GABA receptor modulators which acutely reduce anxious arousal but result in tolerance and side effects when used chronically. Several novel pharmacotherapies (either FDA-approved for other indications or currently in development) may chronically normalize deficient GABA signaling without the downsides of chronic benzodiazepines. Given heterogeneity in PTSD, precision phenotyping will be critical for assigning these treatments to Veterans most likely to benefit, i.e. to an HA-PTSD group with deficient GABA signaling. The investigators propose that RAMP dynamic inhibition can serve as a specific, objective phenotypic target for positive GABA modulation in HA-PTSD. While preliminary data from the investigators has established a specific relationship between dynamic inhibition and fear (relative to negative affect), a crucial step prior to clinical use is validation of the relationship between dynamic inhibition and GABA receptor modulation. The investigators propose to test this causal relationship using the benzodiazepine lorazepam as a pharmacologic probe (rather than a clinical treatment). The validated phenotypic target can then be used for subgroup assignment and mechanistic outcome-tracking in trials of novel GABAergic agents for HA-PTSD.

The investigators hypothesize that the HA-PTSD group will show greater enhancement in dynamic inhibition than other groups with lorazepam compared to placebo. To test this hypothesis, the investigators propose a randomized crossover study in which HA-PTSD, LA-PTSD, and HC Veterans receive a single dose of the lorazepam and placebo in separate experimental sessions in which they perform the RAMP paradigm. Research suggests that arousal-related neural regions may specifically mediate the benefits of GABAergic modulation in HA-PTSD, which could enable targeting of more specific GABAergic treatments. The investigators will therefore examine specific neural mechanisms of GABAergic modulation using fMRI combined with dynamic inhibition as a phenotypic marker.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

1. Veteran;
2. 18-65 years of age, inclusive;
3. Participants must be willing to abstain from alcohol 24 hours prior to and 24 hours after the testing session;
4. Participants must be able to participate and willing to give written informed consent and to comply with the study restrictions;

Additional Inclusion Criteria for PTSD Group:

(a) Current diagnosis of PTSD based on CAPS-5.

Exclusion Criteria:

Exclusion Criteria:

1. Has uncontrolled, clinically significant neurologic (including seizure disorders), cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, immunologic, endocrine disease, or psychiatric disorder, or other abnormality, which may impact the ability of the subject to participate or potentially confound the study results;
2. Pregnancy (assessed by urine test at time of screening and prior to administration of study medication) or lactation;
3. Lifetime history of a chronic psychotic disorder or bipolar disorder type I as assessed by MINI;
4. Current moderate or severe substance use disorder as assessed by MINI;
5. Positive urine toxicology (drugs of abuse as determined by a positive urine test) at screening and before drug administration. Subjects who screen positive for THC will be given an opportunity to be included in the event of a negative urine test 2 weeks later. THC is not infrequently used for medicinal purposes and, in California, is legal for recreational use. Subjects who are positive for THC will therefore not be excluded, but will be retested to ensure that THC is unlikely to be influencing results;
6. Self-report or observable signs of drug or alcohol intoxication or withdrawal;
7. Current benzodiazepine or opioid use; other psychotropic medications are allowed as long as they are at a stable dose for at least 2 weeks and do not exhibit an unsafe interaction with the study medication;
8. Current or recent use of any medication deemed by the study physician (Dr. Howlett) to exhibit an unsafe interaction with lorazepam;
9. Past intolerance (including allergic) to lorazepam or another benzodiazepine;
10. Active suicidal ideation or otherwise considered at high suicidal risk by trained study staff using the C-SSRS;
11. History of a traumatic brain injury (TBI) resulting in loss of consciousness for more than 30 minutes;
12. Volunteers who do not have sufficient command of the English language, or who have any other impairment that would prevent them from reading and understanding the informed consent form(s) and completing the study procedures including clinical testing;
13. Any other reason why, per study physician, the subject should not participate in this study, including concomitant disease or condition that could interfere with, or for which the study drug might interfere with, the conduct of the study, or that would, in the opinion of the study physician, pose an unacceptable risk to the subject in this study.

Additional Exclusion Criteria for HC Group:

(a) Axis I disorder as assessed by MINI.

Additional Exclusion Criteria for fMRI Participants:

1. Contraindication to magnetic resonance imaging.
2. Not right-handed as assessed by Edinburgh Handedness Inventory.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Dynamic inhibition during sensorimotor control | 1.5 hours after dosing
  A dynamic inhibition parameter will be computed for each participant and session using a proportional-derivative (PD) model of sensorimotor control performance on the rapid assessment of motor processing (RAMP) task.

SECONDARY OUTCOMES:
Neural activity during sensorimotor control | 1.5 hours after dosing
  Blood oxygen level dependent (BOLD) response in the dorsal anterior cingulate cortex (dACC), insula, and amygdala (defined according to the Harvard-Oxford anatomical atlas) and in the whole brain will be measured during sensorimotor control performance on the rapid assessment of motor processing (RAMP) task. Bonferroni corrections will be performed based on the number of regions-of-interest (ROIs).
Change from baseline in the the Positive and Negative Affect Schedule - Expanded Form (PANAS X) Fear score | Baseline, 1.5 hours after dosing
  The change from baseline in the PANAS X Fear score will be measured. The PANAS X Fear subscale consists of 6 items. Items are answered on a 5 point scale, 1 (very slightly or not at all) to 5 (extremely). PANAS X Fear scores range from 6-30, with higher scores representing higher levels of fear.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan R Howlett, MD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset will be created and shared. Requests for access must be made in writing signed by a requestor from the United States and include an email address for delivery and an assurance that the recipient will not attempt to identify or re-identify any individual. The request should reference the publication underlying the request. Request may be made to the Principal Investigator/lead point-of-contact for the publication. If the investigator leaves the VA San Diego Healthcare System the requests may be sent to the Associate Chief of Staff for Research.